CLINICAL TRIAL: NCT00842634
Title: A Phase I Study of Autologous T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases SB-728 in HIV-Infected Patients
Brief Title: Autologous T-Cells Genetically Modified at the CCR5 Gene by Zinc Finger Nucleases SB-728 for HIV
Acronym: Zinc-Finger
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Sangamo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 806383
Record Dates: First submitted 2009-02-04; First posted 2009-02-12 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: HIV; HIV Infections
Keywords: HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Patients who have failed two more HAART regimens
  Interventions: Biological: ZFN modified T cells
- Cohort 2 (Experimental): Patients doing well on a stable antiretroviral medication
  Interventions: Biological: ZFN modified T cells; Other: Structured Treatment Interruption
- Cohort 3 (Experimental): Patients who have an undetectable viral load on HAART who have exhibited suboptimal CD4+ T cell gains during long term antiretroviral therapy. This group will not participate in the structured treatment interruption.
  Interventions: Biological: ZFN modified T cells

INTERVENTIONS:
Biological: ZFN modified T cells — A single infusion of 5-10 billion ZFN Modified CD4+ T Cells
Other: Structured Treatment Interruption — Stop Taking HAART Medication for up to 12 weeks (4 weeks after infusion to 16 weeks after infusion)
  Arms: Cohort 2

SUMMARY:
This research study is being carried out to study a new way to possibly treat HIV. This agent is called a "Zinc Finger Nuclease" or ZFN for short. ZFNs are proteins that can delete another protein named CCR5. This CCR5 protein is required for certain common types of HIV (CCR5 tropic) to enter into and infect T-cells. T-cells are one of the white blood cells used by the body to fight HIV. The most important T-cells are those called "CD4 T-cells."

Some people are born without CCR5 on their T-cells. These people remain healthy and are resistant to infection with HIV. Other people have a low number of CCR5 on their T-cells, and their HIV disease is less severe and is slower to cause disease (AIDS).

In order to delete the CCR5 protein on the T cells, this study will isolate large numbers of T-cells from subjects, and then deliver the ZFNs using a delivery vehicle called a viral vector. The viral vector used in this study is called an adenoviral vector. The vector is added to the cells at the beginning of the manufacture process and the ZFNs knock out the CCR5 protein. By the time T-cells are returned to subjects, there is minimal adenovirus or ZFN present. The removal of the CCR5 protein on the T-cells subjects receive, however, is permanent.

The purpose of this research study is to find out whether "zinc finger" modified T-cells are

1. safe to give to humans and
2. find how "zinc finger" modified T cell affects HIV

This is an experimental study. Laboratory studies have shown that when CD4 T-cells are modified with "zinc fingers", HIV is prevented from killing the CD4 T cells. On the basis of these laboratory results, there is the potential that "zinc fingers" may work in humans infected with HIV and improve their immune system by allowing their CD4 T-cells to survive longer (HIV usually kills T cells it infects).

All subjects who receive ZFN Modified CD4+T cells will enroll in a Long Term, Follow-up study to monitor subjects. Subjects will be followed every 3 months for four years. If the ZFN Modified CD4+T cells are no longer found in the blood after four years, then subjects will be contacted yearly for the next 6 years. If the ZFN Modified CD4+T cells are found in the blood at year four, then the subjects will continue to be seen once a year until the ZFN Modified CD4+T cells are no longer found in the blood for a maximum of 10 years.

DETAILED DESCRIPTION:
Cohort 1 - Patients who have failed two more HAART regimens (6 subjects)

Cohort 2 - Patients doing well on a stable antiretroviral medication (6 subjects)

Cohort 3 - Patients who have an undetectable viral load on HAART who have exhibited suboptimal CD4+ T cell gains during long term antiretroviral therapy. This group will not participate in the structured treatment interruption. (6 subjects)

1. Eligibility: Physical Exam, Medical History, Blood Draws for clinical labs and research.
2. 1st Procedure to collect T cells (called apheresis)
3. 2nd Procedure to collect T cells (called apheresis occurs ~3 weeks after 1st Apheresis)and Rectal Biopsy
4. Clinic visit: Physical Exam, Blood Draw for clinical labs and research (~1 to 2 weeks after 2nd Apheresis)
5. Infusion of ZFN modified T cells (~2weeks after Clinic Visit)

   Cohort 1 and Cohort 3 only:
6. Follow up Clinic Visits 48, 72 hours; 1,2,3,6 weeks; 2,3,6, 9 months after ZFN infusion.

Cohort 2 Only:

6. Stop Antiretroviral Medications 4 Weeks after ZFN modified T cell Infusion.

7. Follow-up Clinic Visits 6, 8, 10, 12, 16, weeks after ZFN modified T cell Infusion.

8. Restart Antiretroviral Medications 20 weeks after ZFN modified T cell Infusion.

9. Follow-up Clinic Visits: monthly visits until no detectable HIV found in blood.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1 Only:

* Patients who have been on two more HAART regimens and have failed due to resistance or tolerance (no changes to treatment within 4 weeks of study entry), and who have no viable treatment options likely to result in complete viral suppression.
* CD4+ T cell count of ≥200 cells/mm3
* HIV-1 RNA ≥2000 copies/mL obtained within 60 days prior to study entry performed with an ultrasensitive HIV-1 PCR assay.
* Two HIV-1 RNA levels <150,000 copies/mL obtained within 60 days prior to study entry performed with an ultrasensitive HIV-1 PCR assay. These HIV-1 RNA measurements must be at least 48 hours apart and may include the HIV-1 RNA measurement done at the time of the screening visit.
* Ongoing treatment with HIV entry inhibitors such as enfurvitide or maraviroc are excluded

Cohort 2 Only:

* On a stable antiretroviral medication (no changes to treatment within 4 weeks of study entry) and be willing to continue on current antiretroviral therapy for the duration of the study until undergoing structured treatment interruption.
* CD4+ T cell count of ≥450 cells/mm3 at screen; and a documented CD4 nadir of not lower than 300 cells/mm.
* HIV-1 RNA undetectable by ultrasensitive HIV PCR assay obtained within 60 days prior to study entry performed with an ultrasensitive HIV-1 PCR assay.

Cohort 3 only:

* On a stable antiretroviral medication (no changes to treatment within 4 weeks of study entry) and be willing to continue on current antiretroviral therapy for the duration of the study.
* CD4+ T cell count that is persistently <500 cells/mm3 despite at least 2 years of stable HAART and >200 cells/mm3 at screen
* Subjects must have received at least 2 continuous years of therapy and have had undetectable viral loads by ultrasensitive assay since 6 months of therapy. Subjects who have had a single viral load blip at any point in this time, or who experience intermittent isolated episodes of detectable low-level viremia (detectable but <1000 copies RNA/mL; blips) will remain eligible.
* Subjects who are currently taking maraviroc or have received maraviroc within 6 months of study entry are excluded.

Inclusion for Cohort 1, Cohort 2, Cohort 3:

* HIV-1 infection, as documented by ELISA and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
* Adequate venous access and no other contraindications for leukapheresis.
* Laboratory values obtained at screen. Hemoglobin: ≥ 10.0 (males); ≥ 9.5 (females) g/dL Absolute neutrophil count (ANC): ≥ 1000/mm3 Platelet count: ≥ 100,000/mm3 Serum creatinine: ≤ 1.5 mg/dL (133µ mol/L) Aspartate aminotransferase (AST) or alanine aminotransferase (ALT): ≤ 2.5 times the upper limit of normal (ULN).
* Subjects must be willing to comply with study-mandated evaluations; including not changing their antiretroviral regimen (unless medically indicated) for 2 months in step 2 (Cohort 1) or until undergoing structured treatment interruption (Cohort 2).
* Karnofsky Performance Score of 70 or higher

Exclusion Criteria:

* Acute or chronic hepatitis B or hepatitis C infection
* Current or prior AIDS diagnosis (Cohort 1 and 2 only)
* History of cancer or malignancy, (basal cell or squamous cell carcinoma of the skin allowed)
* History or problems with uncontrolled heart disease, bleeding or hemodynamic instability.
* Have been previously treated with any HIV experimental vaccine within 6 months prior to screening, or any previous gene therapy using an integrating vector.
* Use of the following medications within the last 30 days: chronic corticosteroids, hydroxyurea, or immunomodulating agents (e.g., interleukin-2, interferon-alpha or gamma, granulocyte colony stimulating factors, etc.)
* Breast-feeding, pregnant, or unwilling to use acceptable methods of birth control.
* Use of aspirin, dyprydamole, warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2-week period prior to leukapheresis.
* Active drug or alcohol use or dependence that in the opinion of the investigator, would interfere with adherence to study requirements
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry.
* Receipt of a vaccination within 30 days prior to study entry.
* Have an allergy or hypersensitivity to study product excipients (human serum albumin, DMSO and Dextran 40).
* Currently taking medications called HIV entry inhibitors such as enfuvirtide or maraviroc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety - Treatment related adverse events | Cohort 1, Cohort 3 approximately 1 year from screening. Cohort 2 approximately 40 weeks from screening

SECONDARY OUTCOMES:
Compare the percent of CD4+ and CD8+ T cells that secrete cytokines as a response to stimulation by HIV-specific antigens after the infusion of αCCR5 ZFN-modified autologous T cells | 8 weeks after the infusion of αCCR5 ZFN-modified autologous T cells
Compare the CD4+ and CD8+ T cells response following stimulation by HIVspecific antigens, at baseline and 8 weeks after the infusion of CCR5 ZFN-modified autologous T cells. | 8 weeks after the infusion of CCR5 ZFN-modified autologous T cells
To evaluate the change between baseline CD4+ T-cell count and the average of two consecutive CD4+ T-cell count values after dosing and just prior to initiation of a new drug regimen or at weeks 8 and 12, whichever comes first. | week 8 or 12
Cohort 1: To evaluate the change between baseline log10 HIV-1 RNA level and the average of two consecutive viral load measurements of log10 HIV-1 RNA levels after dosing. | weeks 8 and 12
Cohort 2: To evaluate the time to recrudescence to >500 copies/ml viral load, and viral set point following STI as defined by the average of week 12 and 16 readings (week 8 and 12 post STI). | Week 8 and Week 12
To examine the persistence of CCR5 ZFN-modified autologous T cells in peripheral blood and gut mucosae. | Cohort 1,3: Week 6 and Month 9. Cohort 2: Day 21, Week 16
To monitor for viral drift from CCR5 to CXCR4 trophic virus post treatment using the Monogram Trofile assay, and change in genotypic viral resistance profile using the Monogram GenSeq assay. | Cohort 2 only: Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Tebas, MD, Principal Investigator — University of Pennsylvania; David Stein, MD, Principal Investigator — Jacobi Medical Center
Locations (2):
- United States (2):
  - Jacobi Medical Cener, The Bronx, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tebas P, Stein D, Tang WW, Frank I, Wang SQ, Lee G, Spratt SK, Surosky RT, Giedlin MA, Nichol G, Holmes MC, Gregory PD, Ando DG, Kalos M, Collman RG, Binder-Scholl G, Plesa G, Hwang WT, Levine BL, June CH. Gene editing of CCR5 in autologous CD4 T cells of persons infected with HIV. N Engl J Med. 2014 Mar 6;370(10):901-10. doi: 10.1056/NEJMoa1300662. PMID 24597865
- See also: Clinical Trials Listing for UPENN HIV Clinical Trials Unit — http://www.uphs.upenn.edu/pennactu/